CLINICAL TRIAL: NCT01984619
Title: A Prospective Study Evaluating the Treatment of Hyperdynamic Forehead Wrinkles Utilizing the Iovera With Blunt Tip Cannula Smart Tip
Brief Title: Prospective Study Evaluating the Treatment of Hyperdynamic Forehead Wrinkles
Status: Completed | Type: Observational
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MYO-0834
Record Dates: First submitted 2013-10-29; First posted 2013-11-15 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Wrinkles
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Blunt Tip Cannula
  Interventions: Device: Cryotherapy for the utilization of wrinkle reduction (iovera)

INTERVENTIONS:
Device: Cryotherapy for the utilization of wrinkle reduction (iovera)
  Other Names: iovera

SUMMARY:
To evaluate the safety and effectiveness of the iovera° device with the blunt tip cannula for the treatment of forehead wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Male or Females 18-65 years of age.
* Forehead wrinkle(s) rating of at least 2 in animation on the 5-point Wrinkle Scale (5WS) which upon physical manipulation of the skin demonstrates a reduction in wrinkle severity.
* Subject has at least a 2 point difference between resting and dynamic forehead wrinkle scores using the 5WS.
* Glabellar wrinkle score of "1" or higher in animation on the 5-point Glabella Scale (5GS).
* Fitzpatrick Skin Type I, II, III, or IV.
* Subject has consented and agreed to participate in all study procedures and visits for the study's duration.
* Subject is in good general health, free of any disease state, or physical condition that might impair evaluation of forehead and/or glabellar wrinkle rating or which, in the Investigator's opinion, exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* Subject has a clotting disorder or coagulopathy that requires use of an anticoagulant and/or antiplatelet therapy (e.g., warfarin, clopidigrel, etc.)
* Subject has used medication or supplements affecting clotting cascade (e.g., aspirin, fish oil, etc.), or non-steroidal anti-inflammatory drugs (NSAIDs, e.g., ibuprofen and naproxen) within seven (7) days prior to administration of the device.
* Subject has had prior surgery that alters the subcutaneous anatomy of the target treatment sites.
* Subject has undergone another surgical cosmetic procedure or botulinum toxin injection at or above the level of the zygoma (cheekbones) within the past six (6) months prior to administration of the device.
* Subject has a resting wrinkle score of "3" or higher on the 5WS.
* Subjects who actively elevate forehead at rest.
* Subject has been treated with fillers in the temple or forehead area in the time intervals specified prior to the start of their participation in the study.
* Subject has any of the following:

  1. Dermatochalasis with <1mm lid margin when looking straight ahead.
  2. Excessive skin laxity.
  3. Asymmetry in the upper face.
  4. History of facial nerve palsy.
  5. Eyebrow or eyelid ptosis.
  6. History of neuromuscular disorder.
  7. Chronic dry eye symptoms.
  8. Allergy or intolerance to local anesthetic agents (e.g., Lidocaine).
  9. Use of narcotic medication for a chronic pain condition.
  10. Any other clinically significant, in the opinion of the Investigator, local skin condition (e.g., skin infection) at target treatment site that may interfere or be a safety concern.
  11. Any physical or psychiatric condition that in the Investigator's opinion would prevent adequate study participation.
  12. Chronic medical condition that in the Investigator's opinion would affect study participation (such as uncontrolled hypertension, diabetes, hepatitis, HIV, etc.).
  13. Diagnosis of:

      * Cryoglobinemia
      * Paroxysmal cold hemoglobinuria
      * Cold Uticaria
      * Raynaud's Disease
      * Open and/or infected wounds
      * Existing neuromuscular disease
  14. Fitzpatrick Skin Type V or IV
  15. Subject is currently enrolled in an investigational drug, biologic or device study that could affect the safety or effectiveness of the iovera° treatment.
  16. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, male or female, age 18 - 65 with forehead wrinkles deemed significant per protocol inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Wrinkle severity when eyebrows are elevated at 30 days post-treatment. | 120 Days

OTHER OUTCOMES:
Anticipated observations, adverse events and SAEs/UADEs will be assessed at each visit. | 120 Days

CONTACTS AND LOCATIONS:
Locations (1):
- The Aesthetics Research Center, Redwood City, California, United States